CLINICAL TRIAL: NCT02166008
Title: Cytoprotective Agent for Peptic Ulcer Prevention in Patients Taking Dual Antiplatelet Agents: A Randomized Double-blind Placebo Control Trial Study
Brief Title: Cytoprotective Agent and Peptic Ulcer in Dual Antiplatelet :RCT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, MD, Doctor, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP006
Record Dates: First submitted 2013-09-30; First posted 2014-06-18 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Gastric Ulcer Induced by Anti-platelet Agent; Duodenal Ulcer Induced by Anti-platelet Agent
Keywords: Repamipide; Dual antiplatelet; Peptic ulcer
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Repamipide (Active Comparator): Rebamipide (100) 1 tab oral tid for 1 year or peptic ulcer occurred
  Interventions: Drug: Repamipide
- placebo (Placebo Comparator): A placebo is a simulated or otherwise medically ineffectual treatment for a disease or other medical condition intended to deceive the recipient. It will be prescribed as the same regimen of Rabamipide.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Repamipide
  Arms: Repamipide
Drug: Placebo
  Other Names: Placebo will be made in the same configuration of rabamipide
  Arms: placebo

SUMMARY:
* Primary objective : To evaluate the efficacy of Rapamide in peptic ulcer prevention in patients taking dual antiplatelet agents
* Study Design: Single center, double-blind, randomized-control trial study
* Study drug: Repamipide vs. placebo
* Assessment criteria The patients will be discharged from the study when one of the followings occurred,

  1. Peptic ulcer from upper endoscopy at 3 and 6 month follow up
  2. Clinical of upper gastrointestinal bleeding with peptic ulcer from upper endoscopy
  3. Anemia by CBC at 1,3 ,6,12 month with peptic ulcer from upper endoscopy
  4. Evidence of recurrent myocardial infarction from stent thrombosis

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 year-old
2. Had cardiovascular disease which needed clopidogrel and aspirin
3. Stable enough for gastroscopy

Exclusion Criteria:

1. Gastroscopy revealed peptic ulcer
2. Had contraindication for gastroscopy
3. Not allowed for gastroscopy by cardiologist

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
number of peptic ulcer by end0scopy | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Patumwan, Bangkok, Thailand

REFERENCES:
- [Derived] Pittayanon R, Piyachaturawat P, Rerknimitr R, Prueksapanich P, Chaitongrat S, Lertsuwunseri V, Srimahachota S, Mahachai V. Cytoprotective agent for peptic ulcer prevention in patients taking dual antiplatelet agents: A randomized, double-blind placebo-controlled trial. J Gastroenterol Hepatol. 2019 Sep;34(9):1517-1522. doi: 10.1111/jgh.14671. Epub 2019 May 8. PMID 30919492
- See also: Institutional review board, Faculty of medicine, Chulalongkorn University — http://www.medchulairb.com